CLINICAL TRIAL: NCT05196620
Title: Prevalence of Anal Sphincter Defects After Childbirth in Primiparous Women
Brief Title: Prevalence of Anal Sphincter Defects After Childbirth
Acronym: PRADA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Hospital Clínico Universitario Lozano Blesa (Other); Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Principal Investigator, Jose-M Ramirez, Prof, Universidad de Zaragoza
Other Study IDs: UZaragoza-3
Record Dates: First submitted 2021-12-29; First posted 2022-01-19 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Fecal Incontinence; Childbirth Problems
Keywords: Anal Ultrasound; Fecal Incontinence; Childbirth
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EAUS: Patients with EAUS pre and postpartum
  Interventions: Other: Endoanal Ultrasound (EAUS)

INTERVENTIONS:
Other: Endoanal Ultrasound (EAUS) — Endoanal Ultrasound pre- and postpartum

SUMMARY:
The incidence of obstetric sphincter tears has risen to 15-30% and the prevalence of anal incontinence (AI) symptoms after childbirth may be as high as 40%. The present study aims to evaluate the prevalence of anal sphincter defects after childbirth in primiparous women-

DETAILED DESCRIPTION:
The incidence of sphincter defect in women has raised in recently with current rates as high as 30% after vaginal deliveries. Fecal incontinence could be present at the time of the delivery but it is a real problem longtime after, in women older than 60 years.

It is of great importance not only an early detection but to indicates the best possible management as soon as posible.

The design is a prospective observational study including primiparous woman, without previous anal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous pregnant patients aged >18 y, evaluated during pregnancy and after childbirth, including both vaginal and cesarean deliveries.

Exclusion Criteria:

* Non primiparous patients and patients with a history of anal surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — It is a study about childbirth problems.
Study Population: Primaparous pregnat
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Integrity of anal sphincter | 4 months
  No defect detected on EAUS
Defects on anal canal | 4 months
  Disruption of any of the anal canal sphincters

SECONDARY OUTCOMES:
QoL | 4 months
  According to a dedicated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jose-M Ramirez, Prof, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Hospital Clinico Lozano Blesa, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tejedor P, Plaza J, Bodega-Quiroga I, Ortega-Lopez M, Garcia-Olmo D, Pastor C. The Role of Three-Dimensional Endoanal Ultrasound on Diagnosis and Classification of Sphincter Defects After Childbirth. J Surg Res. 2019 Dec;244:382-388. doi: 10.1016/j.jss.2019.06.080. Epub 2019 Jul 17. PMID 31325659
- [Background] Sultan AH, Thakar R. Diagnosis of anal sphincter tears to prevent fecal incontinence: a randomized controlled trial. Obstet Gynecol. 2005 Nov;106(5 Pt 1):1108-9; author reply 1109. doi: 10.1097/01.AOG.0000186051.88740.7f. No abstract available. PMID 16260538
- [Background] Johannessen HH, Wibe A, Stordahl A, Sandvik L, Morkved S. Do pelvic floor muscle exercises reduce postpartum anal incontinence? A randomised controlled trial. BJOG. 2017 Mar;124(4):686-694. doi: 10.1111/1471-0528.14145. Epub 2016 Jun 7. PMID 27272501
- [Background] Damon H, Bretones S, Henry L, Mellier G, Mion F. Long-term consequences of first vaginal delivery-induced anal sphincter defect. Dis Colon Rectum. 2005 Sep;48(9):1772-6. doi: 10.1007/s10350-005-0075-z. PMID 15981061
- [Background] Harvey MA, Pierce M, Alter JE, Chou Q, Diamond P, Epp A, Geoffrion R, Harvey MA, Larochelle A, Maslow K, Neustaedter G, Pascali D, Pierce M, Schulz J, Wilkie D, Sultan A, Thakar R; Society of Obstetricians and Gynaecologists of Canada. Obstetrical Anal Sphincter Injuries (OASIS): Prevention, Recognition, and Repair. J Obstet Gynaecol Can. 2015 Dec;37(12):1131-48. doi: 10.1016/s1701-2163(16)30081-0. PMID 26637088
- [Background] Thomas GP, Gould LE, Casunuran F, Kumar DA. A retrospective review of 1495 patients with obstetric anal sphincter injuries referred for assessment of function and endoanal ultrasonography. Int J Colorectal Dis. 2017 Sep;32(9):1321-1325. doi: 10.1007/s00384-017-2851-3. Epub 2017 Jul 7. PMID 28685224